CLINICAL TRIAL: NCT03624361
Title: A Prospective, Open, Multicentre Clinical Trial With One Cohort Analysing the Efficacy and Safety of MINIject in European Patients With Open Angle Glaucoma Uncontrolled by Topical Hypotensive Medications
Brief Title: MINIject Glaucoma Implant in European Patients
Acronym: STAR-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: iSTAR Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STAR-II (ISM04EU)
Record Dates: First submitted 2018-05-28; First posted 2018-08-10 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Glaucoma, Open-Angle; Glaucoma Eye; Intraocular Pressure
Keywords: Minimally Invasive Glaucoma Surgery; Glaucoma Implant; Lower IOP; IOP; Intraocular Pressure
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Intervention Model Description: MINIject glaucoma implant CS600 with Dual Operator Delivery Tool
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stand-alone (Experimental): Patients will receive MINIject Glaucoma implant in a stand-alone procedure.
  MINIject implant is used to reduce intra-ocular pressure in the eye through a minimally-invasive Glaucoma surgical intervention.
  Interventions: Device: Glaucoma device implantation in a stand-alone procedure

INTERVENTIONS:
Device: Glaucoma device implantation in a stand-alone procedure — MINIject implant is used to reduce intra-ocular pressure in the eye through a minimally-invasive Glaucoma surgical intervention.
  The intervention is to be performed as stand-alone surgery.

SUMMARY:
The study will evaluate the efficacy and safety of the MINIject glaucoma implant and Intraocular Pressure (IOP) lowering effects with or without glaucoma medications. The procedure will be a stand-alone surgery. Overall, the patient will be asked to perform several examinations up to 24 months after surgery.

DETAILED DESCRIPTION:
The primary endpoint is the 'qualified success' rate at 6 months after surgery greater than 60%. 'Qualified success' is defined as a diurnal IOP ≤ 21mmHg (millimeter mercury) and > 5mmHg with a minimum 20% diurnal IOP reduction from baseline with or without the concomitant use of allowed glaucoma hypotensive medication at 6 months after surgery

ELIGIBILITY:
Inclusion Criteria:

* Males or females, 50 years of age or older.
* Diagnosis of primary open angle glaucoma during screening visit or earlier.
* Grade 3 (open, 20-35 degrees) or grade 4 (wide open, 35-45 degrees) according to Shafer Angle Grading System.

Exclusion Criteria:

* Diagnosis of glaucoma other than primary open angle glaucoma (e.g. angle closure glaucoma or secondary open angle glaucoma) in the study eye.
* Grade 2 (narrow, 20 degrees), grade 1 (extremely narrow, less or equal to 10 degrees) and grade 0 (closed or slit) according to Shafer Angle Grading System.
* Neovascular glaucoma in the study eye.
* Corneal opacity or iridocorneal angle not visible through gonioscopy prisma in the study eye, preventing correct placement of the implant.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Qualified success for lowering the IOP | at 6 months
  The primary objective is the 'qualified success' rate at 6 months after surgery greater than 60%. 'Qualified success' is defined as a diurnal IOP ≤ 21 mmHg and > 5 mmHg with a minimum 20% diurnal IOP reduction from baseline with or without the concomitant use of allowed glaucoma hypotensive medication at 6 months after surgery

SECONDARY OUTCOMES:
Safety assessment of device in terms of adverse events (AEs) and serious adverse events (SAEs) reported during duration of study | up to 24 months after surgery
  show safety of the MINIject implant and the procedure used to implant the device

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Pfeiffer, Prof., Principal Investigator — Universitätsklinikum Mainz
Locations (8):
- France (2):
  - Center Hospotalier Universitaire Genoble Alpes, Grenoble
  - Hôpital de la Croix Rousse, Lyon
- Germany (5):
  - Ludwig-Maximilians-University Munich, Munich, Bavaria
  - Uni-Augenklinik Bochum, Bochum, North Rhine-Westphalia
  - Uniklinik Köln, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Mainz, Mainz, Rhineland-Palatinate
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
- Hospital Clínico San Carlos, Madrid, Spain

REFERENCES:
- [Result] Garcia Feijoo J, Denis P, Hirneiss C, Aptel F, Perucho Gonzalez L, Hussain Z, Lorenz K, Pfeiffer N; STAR-II Investigators. A European Study of the Performance and Safety of MINIject in Patients With Medically Uncontrolled Open-angle Glaucoma (STAR-II). J Glaucoma. 2020 Oct;29(10):864-871. doi: 10.1097/IJG.0000000000001632. PMID 32769736
- See also: Homepage of the company and information about the product — https://www.istarmed.com/